CLINICAL TRIAL: NCT00441662
Title: Sub-Tenon Triamcinolone in the Prevention of Radiation-Induced Macular Edema Following Plaque Radiotherapy for Uveal Melanoma
Brief Title: Sub-Tenon Triamcinolone in the Prevention of Radiation-Induced Macular Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Wills Eye Sub-Tenon Kenalog
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Melanoma
Keywords: Melanoma; Uvea; Macula; Edema; Plaque radiotherapy; Brachytherapy; Triamcinolone
MeSH Terms: conditions — Melanoma; Edema

INTERVENTIONS:
Drug: Sub-Tenon triamcinolone 40mg

SUMMARY:
Melanoma is the most common primary tumour which occurs inside the eye. For over 20-years, it has been possible, in many cases, to use local delivery of radiation to the eye to treat this type of tumour, avoiding the need to surgically remove the affected eye. This treatment, however, is often complicated by radiation-induced loss of vision, months or years after treatment.

The aim of this research project is to investigate the potential prevention of radiation complications in the eye by giving anti-inflammatory medication (a long-acting steroid) in the form of a local injection around the eye at the time of treatment, and at 4-months and 8-months following treatment. This medication (named 'triamcinolone') has been successfully used to treat similar complications of diabetic eye disease, for example, and has a good safety profile.

The rationale of this study is to attempt to preserve vision, in addition to preserving the eye, in patients affected by this eye tumour, and therefore preserve quality of life for these patients.

DETAILED DESCRIPTION:
BACKGROUND: Uveal melanoma is the most common primary intraocular malignancy. Plaque radiation (brachytherapy) has emerged as the most common treatment in the current management of uveal melanoma, but is complicated by visual loss in close to 70% of patients at 10 years follow-up. Strategies for the prevention and early treatment of radiation retinopathy (and radiation maculopathy in particular) need to be developed to improve visual outcome following eye-conserving treatment of uveal melanoma. Triamcinolone, a long acting locally-administered corticosteroid, is of established benefit in macular oedema from other causes.

PURPOSE: This study will evaluate the efficacy of sub-Tenon triamcinolone in the prevention of radiation maculopathy in patients undergoing plaque radiotherapy for uveal melanoma.

DESIGN: A prospective randomised control study.

STUDY POPULATION: 170 patients undergoing plaque radiation treatment for uveal melanoma.

SETTING: Ocular Oncology Service, Wills Eye Hospital, Philadelphia, USA.

INTERVENTION: Triamcinolone acetonide (40 mg in 1 cc) injected into the sub-Tenon space using sterile technique at the time of plaque radiotherapy and 4 and 8 months later.

OUTCOME MEASURES: Visual acuity, optical coherence tomographic (OCT) analysis of macular architecture and foveal thickness, at 4, 8, and 12 months following brachytherapy.

EXCLUSION CRITERIA: Pre-existing macular disease (e.g. age-related macular degeneration, diabetic maculopathy, vascular occlusion, macular hole); prior retinal detachment; media opacities precluding accurate OCT imaging; history of intraocular pressure elevation related to corticosteroid treatment -'steroid responder'; history of glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Uveal melanoma new diagnosis, undergoing plaque radiation treatment

Exclusion Criteria:

* Pre-existing macular disease
* age-related macular degeneration
* diabetic maculopathy
* pre-existing retinal vascular occlusion
* macular hole
* surface wrinkling retinopathy
* prior retinal detachment
* media opacities precluding accurate OCT imaging
* known 'steroid responder'
* glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170
Dates: Start 2004-11; Study Completion 2007-05

PRIMARY OUTCOMES:
Presence of macular edema on optical coherence tomography

SECONDARY OUTCOMES:
Grade of macular edema on optical coherence tomography
Foveal thickness measurement by optical coherence tomography
Visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Carol L Shields, M.D., Principal Investigator — Ocular Oncology Service, Wills Eye Institute
Locations (1):
- Ocular Oncology Service, Wills Eye Institute, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Shields CL, Shields JA, Gunduz K, Freire JE, Mercado G. Radiation therapy for uveal malignant melanoma. Ophthalmic Surg Lasers. 1998 May;29(5):397-409. PMID 9599365
- [Background] Shields CL, Shields JA, Cater J, Gunduz K, Miyamoto C, Micaily B, Brady LW. Plaque radiotherapy for uveal melanoma: long-term visual outcome in 1106 consecutive patients. Arch Ophthalmol. 2000 Sep;118(9):1219-28. doi: 10.1001/archopht.118.9.1219. PMID 10980767
- [Background] Shields CL, Cater J, Shields JA, Chao A, Krema H, Materin M, Brady LW. Combined plaque radiotherapy and transpupillary thermotherapy for choroidal melanoma: tumor control and treatment complications in 270 consecutive patients. Arch Ophthalmol. 2002 Jul;120(7):933-40. doi: 10.1001/archopht.120.7.933. PMID 12096964
- See also: Related Info — http://www.etrf.org
- See also: Related Info — http://www.eyecancerbook.com